CLINICAL TRIAL: NCT06271356
Title: Effect of a Navigation Intervention on Care Equity for Women of Color Diagnosed With Breast Cancer: A Feasibility Study
Brief Title: Breast Cancer - Navigate - Prospective Cohort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: The Chrysalis Initiative (Unknown)
Responsible Party: Principal Investigator, Betina Yanez, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00220278
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Quality of Life; Chemotherapy
Keywords: eHealth
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BC-Navi (Experimental): Apply TCI's patient navigation-and-coaching program and its website/mobile app (Breast Cancer-Navigate) platform to improve timely initiation to patient adjuvant chemotherapy treatment among diverse breast cancer patients.
  Interventions: Behavioral: BC-Navigate

INTERVENTIONS:
Behavioral: BC-Navigate — BC-Navigate is a website/application to help guide women through care delivery during breast cancer treatment.

SUMMARY:
The Chrysalis Initiative (TCI) has with its technology partner Eversana/Intouch developed the BC-Navigate website/application to help guide women through care delivery during breast cancer treatment.

TCI a nonprofit, breast cancer education and navigation organization is developing methods to address health inequities in cancer care delivery. TCI and its new academic/clinical partner, The Robert H. Lurie Comprehensive Cancer Center of Northwestern University, propose to apply TCI's developed patient navigation support techniques to enhance knowledge and self-advocacy among a cohort of Black and African American women, and other women of color (WOC), receiving care in Northwestern's breast cancer program.

Therefore, the purpose of this study is to apply TCI's patient navigation-and-coaching program and its website/mobile app (Breast Cancer-Navigate) platform to improve timely initiation to patient adjuvant treatment among WOC breast cancer patients and evaluate the feasibility and preliminary efficacy of this approach.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Diagnosed with non-metastatic breast cancer (stages I-III)
* An order placed for a post-operative chemotherapy cycle by a NM clinician
* Not have initiated a recommended post-operative chemotherapy cycle at the time of study enrollment
* Completed surgery for breast cancer
* First-time diagnosis of breast cancer
* Established care at Northwestern Medicine
* English-speaking as the navigation website is not yet available in other languages
* Access to internet on a smart phone or computer/tablet
* Any ethnic background
* We will only consider patients that sign an informed consent form

Exclusion Criteria:

* Men will be excluded because the navigation website only contains content and resources for women. Men also make up less than 1% of all breast cancer diagnoses and the Breast Cancer-Navigate app/website content was developed for female breast cancer patients.
* Diagnosis of additional, life-threatening condition (e.g., end-stage renal disease, heart failure) which can interfere with timely planned adjuvant chemotherapy treatment for cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Demand of BC-Navi: Recruitment Rate | 12 weeks
  We assess the demand for the BC-Navi application through study recruitment. Based on previous psychosocial and behavioral studies in oncology, a 75% recruitment rate is considered adequate.
Demand of BC-Navi: Retention Rate | 12 weeks
  Another way we assess demand of the BC-Navi application is through participant retention. Based on previous psychosocial and behavioral studies in oncology, a 75% retention rate is considered adequate .
Acceptability of BC-Navi | 12 weeks
  To assess acceptability, all participants are asked to complete an exit interview on BC-Navi. This interview assesses the usefulness, satisfaction, learnability, and usability of the application. This exit interview was synthesized from validated measures assessing eHealth intervention acceptability, and was adapted for our study to better fit our target population and our application design. Above-average scores on the questionnaire are considered acceptable.
Preliminary Efficacy: Chemotherapy Initiation | 12 weeks
  Preliminary efficacy will be measured by time to chemotherapy initiation, which will be operationalized as chemotherapy treatment initiation within 90 days of completion of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No